CLINICAL TRIAL: NCT02490696
Title: Comparative Study of the Hypoxia Measured in FAZA and F-miso TEP/CT Scan in Patients With Non-small Cell Lung Cancer at the Time of Diagnosis : Correlation With Immunohistochemistry
Brief Title: Comparative Study of the Hypoxia Measured in FAZA and F-miso PET/CT Scan in Patients With Non-small Cell Lung Cancer
Acronym: RTEP6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHB14.01
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PET scan; FAZA; F-Miso; hypoxia; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hypoxia; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miso (Experimental): In this arm two PET scans wiil be realized. The first one will be made with F-Miso tracer. 24 hours later the FAZA PET scan will be performed. 24 hours after the last PET scan the surgery will be realized. During this surgery a piece of tumor will be collected and analyse by immunohistochemistry for markers of hypoxia
  Interventions: Device: Miso PET scan
- FAZA (Experimental): In this arm two PET scans wiil be realized. The first one will be made with FAZA tracer. 24 hours later the F-Miso PET scan will be performed. 24 hours after the last PET scan the surgery will be realized. During this surgery a piece of tumor will be collected and analyse by immunohistochemistry for markers of hypoxia
  Interventions: Device: FAZA PET scan

INTERVENTIONS:
Device: Miso PET scan — 2 PET scans will be performed before surgery : the first one with F-Miso tracer and the second, 24 hours later, with FAZA tracer
  Arms: Miso
Device: FAZA PET scan — 2 PET scans will be performed before surgery : the first one with FAZA tracer and the second, 24 hours later, with F-Miso tracer
  Arms: FAZA

SUMMARY:
The purpose of the study is to compare the intratumoral biodistribution of FAZA and F-miso in patients with non-small cell lung cancer and correlate the results of PET scans with immunohistochemistry.

DETAILED DESCRIPTION:
The aim of the study is to compare the biodistribution of the two tracers specific for hypoxia in patients with non-small cell lung cancer.

Two PET scans will be performed with FAZA and F-Miso tracers. The time between these twi PET scans will be 24 hours.

another 24 hours after the late PET scan, the surgery will be done and a piece of tumor will be collected.

Piece of tumor will be analysed by immunohistochemistry for hypoxia markers.

The results of immunohistochemistry will be correlated with the biodistribution of the two tracers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* More than 18 years old
* Patient with non-small cell lung cancer (histologically proved)
* PS inferior or equal to 1 (good general state)
* Patient must have surgery for their non-small cell lung cancer
* Stage of tumor Superior or equal to 2a without metastasis
* Tumoral fixation with 18-FDG-PET superior to mediastinal background noise
* Written inform consent

Exclusion Criteria:

* Histology other than primitive non-small cell lung cancer
* In situ form at the histological study
* Patient without evaluable target
* No fixation on the pretherapeutic FDG-PET scan
* PS Superior or equal to 2
* neoplastic disease (less than 2 years or progressive)
* Pregnant woman or child-bearing
* Patient Under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Comparison of hypoxia with FAZA and F-Miso tracer | one year
  SUV max, SUV mean and SUV peak were calculated for FAZA PET and Fmiso PET and will be correlated with results of immunohistochemistry

SECONDARY OUTCOMES:
overall survival | one year
  time between inclusion and the death whatever the cause
disease-free survival | one year
  time between inclusion and the progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vera, MD, PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Texte E, Gouel P, Thureau S, Lequesne J, Barres B, Edet-Sanson A, Decazes P, Vera P, Hapdey S. Impact of the Bayesian penalized likelihood algorithm (Q.Clear(R)) in comparison with the OSEM reconstruction on low contrast PET hypoxic images. EJNMMI Phys. 2020 May 12;7(1):28. doi: 10.1186/s40658-020-00300-3. PMID 32399752